CLINICAL TRIAL: NCT07170059
Title: An Observational Study on the Impact of Herpes Zoster Vaccine on the Incidence of Herpes Zoster and Survival in Lung Cancer Patients
Brief Title: Observational Study on the Impact of Herpes Zoster Vaccine on the Incidence of Herpes Zoster and Survival in Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yalei Zhang, The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: ZSHV-LC-OBS2025
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccination group: Lung cancer patients receive herpes zoster vaccine
  Interventions: Biological: herpes zoster vaccine
- Unvaccinated group: Lung cancer patients have not received herpes zoster vaccine

INTERVENTIONS:
Biological: herpes zoster vaccine — Receive the herpes zoster vaccine; Do not receive the herpes zoster vaccine
  Groups: Vaccination group

SUMMARY:
To evaluate the impact of herpes zoster vaccine on the incidence of herpes zoster and survival in lung cancer patients, and to explore its preventive effect and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female patients >=18 years of age; 2.Histological diagnosis of NSCLC, including both non-small cell lung cancer and small cell lung cancer, regardless of whether they are in the early, locally advanced stage or advanced stage, and regardless of whether they have received surgery, radiotherapy, chemotherapy or other treatments; 3. Never received herpes zoster vaccine

Exclusion Criteria:

* Patients having other factors that preventing researchers from enrollment them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients can receive or not receive the herpes zoster vaccine
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of herpes zoster at 12 months | 12 months
  During the 12-month follow-up period, the incidence of herpes zoster in lung cancer patients was evaluated through regular clinical examinations, imaging tests, and laboratory tests.
Incidence of herpes zoster | 24 months
  The proportion of lung cancer patients who developed herpes zoster during the study period.

SECONDARY OUTCOMES:
Survival rate | 5 years
  The survival rate of lung cancer patients within a specific time period (such as 1 year, 2 years, or 5 years).

OTHER OUTCOMES:
Lung cancer-related complications | 5 years
  Severity of herpes zoster and incidence of complications (e.g., postherpetic neuralgia)
Length of hospital stay | 5 years
  Record the number of days of hospitalization for patients hospitalized due to herpes zoster
Hospitalization rate | 5 years
  The proportion of patients hospitalized due to herpes zoster or other related complications.
Immune response | 5 years
  The immune response (such as antibody levels) of patients after vaccination is evaluated through serological testing.
Adverse reactions after vaccination | 30 days
  Observe whether patients who receive the herpes zoster vaccine experience adverse reactions after vaccination, such as fever, redness, swelling and pain at the injection site, headache, dizziness, etc.